CLINICAL TRIAL: NCT00339495
Title: Prostate Lung Colorectal and Ovarian (PLCO) Cancer Screening Trial
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997041; OH97-C-N041
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-02

CONDITIONS: Cancer; Death
Keywords: Prostate; Screening Trial; Ovarian; Lung; Colorectal
MeSH Terms: conditions — Neoplasms; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Screening: Participants received their usual care
- Screening: Participants received trial-provided screening examinations for prostate, lung, colorectal, and ovarian cancer

SUMMARY:
The Division of Cancer Preventionl (DCP, formerly DCPC), under extramural contracts to 10 U.S. clinical centers, is evaluating the effectiveness of screening for prostate, lung, colorectal and ovarian cancer (The PLCO Trial). In 1996 the NCI Executive Committee approved the expansion of the PLCO Trial to collect additional materials and to conduct additional studies. About, 74,000 men and 74,000 women, aged 55-74 years, have been randomized on a 50/50 basis into screening or usual care arms. Additional blood is collected from screened subjects and saliva for buccal cells from control subjects. Pathologic tissues are obtained for selected cases that develop cancer or selected related diseases (e.g. colon polyps, benign prostatic hyperplasia). Additional questionnaire-based risk and disease-related information is also collected, withconfirmation of disease status from medical records. Genetic, biochemical and questionnairebasedrisk information will be related to the development of cancer and other diseases in this population. Volunteers who provide samples for these studies will not routinely receive their individual results from the Additional Investigation. Subjects requesting such information, however, will be provided their test results. In 2009 the NCI Executive Committee approved the Extended Follow-up of subjects beyond the original 13-year follow-up period. Participants will be reconsented for the release of records to a single NCI-Designated Central Data Collection Center (CDCC), which will administer the annual mailings containing the annual study update questionnaire and a brief (1-2 page) risk factor questionnaire. Individuals who do not consent to release their identifiers to the CDCC will be followed up passively through linkage to state cancer registries and the National Death Index.

This protocol Review Application is for (1) the collaboration of intramural scientists in the Division of Cancer Epidemiology and Genetics (DCEG) in the Additional Studies and (2) the coordination, in collaboration with DCP, of the Extended Follow-up.

DETAILED DESCRIPTION:
The Division of Cancer Preventionl (DCP, formerly DCPC), under extramural contracts to 10 U.S. clinical centers, is evaluating the effectiveness of screening for prostate, lung, colorectal and ovarian cancer (The PLCO Trial). In 1996 the NCI Executive Committee approved the expansion of the PLCO Trial to collect additional materials and to conduct additional studies. About, 74,000 men and 74,000 women, aged 55-74 years, have been randomized on a 50/50 basis into screening or usual care arms. Additional blood is collected from screened subjects and saliva for buccal cells from control subjects. Pathologic tissues are obtained for selected cases that develop cancer or selected related diseases (e.g. colon polyps, benign prostatic hyperplasia). Additional questionnaire-based risk and disease-related information is also collected, with confirmation of disease status from medical records. Genetic, biochemical and questionnaire-based risk information will be related to the development of cancer and other diseases in this population. Volunteers who provide samples for these studies will not routinely receive their individual results from the Additional Investigation. Subjects requesting such information, however, will be provided their test results. In 2009 the NCI Executive Committee approved the Extended Follow-up of subjects beyond the original 13-year follow-up period. Participants will be reconsented for the release of records to a single NCI-Designated Central Data Collection Center (CDCC), which will administer the annual mailings containing the annual study update questionnaire and a brief (1-2 page) risk factor questionnaire. Individuals who do not consent to release their identifiers to the CDCC will be followed up passively through linkage to state cancer registries and the National Death Index.

This protocol Review Application is for (1) the collaboration of intramural scientists in the Division of Cancer Epidemiology and Genetics (DCEG) in the Additional Studies and (2) the coordination, in collaboration with DCP, of the Extended Follow-up.

ELIGIBILITY:
* INCLUSION CRITERIA:

Men and women aged 55-74 years who do not have a prior history of PLCO tumors and have not undergone routine screening.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community samples from ten US screening centers: Birmingham AL, Denver CO, Detroit MI, Honolulu HI, Marshfield WI, Minneapolis MN, Pittsburgh PA, Salt Lake City UT, St Louis MO, and Washington DC
Sampling Method: Probability Sample
Enrollment: 154900 (Actual)
Dates: Start 1998-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | Extended beyond T13
  Death
Cancer incidence | Extended beyond T13
  Cancer Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Moore, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Westat, Inc., Rockville, Maryland, United States

REFERENCES:
- [Derived] Malcomson FC, Shams-White MM, Reedy J, Huang WY, Moore SC, Loftfield E. Adherence to the 2018 World Cancer Research Fund/American Institute for Cancer Research Cancer Prevention Recommendations and risk of lifestyle-related cancers in the prostate, lung, colorectal, and ovarian cancer screening trial. BJC Rep. 2025 Nov 19;3(1):81. doi: 10.1038/s44276-025-00195-6. PMID 41261199
- [Derived] Wei W, Wang S, Yuan Z, Ren Y, Wu J, Gao X, Wang R, Li J. Plant-based diets and the risk of lung cancer: a large prospective cohort study. Eur J Nutr. 2025 Feb 1;64(2):73. doi: 10.1007/s00394-024-03570-0. PMID 39891747
- [Derived] Jiang Y, Xie Q, Chen R. Breast Cancer Incidence and Mortality in Relation to Hormone Replacement Therapy Use Among Postmenopausal Women: Results From a Prospective Cohort Study. Clin Breast Cancer. 2022 Feb;22(2):e206-e213. doi: 10.1016/j.clbc.2021.06.010. Epub 2021 Jun 26. PMID 34548240
- [Derived] Wang K, Wu Q, Li Z, Reger MK, Xiong Y, Zhong G, Li Q, Zhang X, Li H, Foukakis T, Xiang T, Zhang J, Ren G. Vitamin K intake and breast cancer incidence and death: results from a prospective cohort study. Clin Nutr. 2021 May;40(5):3370-3378. doi: 10.1016/j.clnu.2020.11.009. Epub 2020 Nov 16. PMID 33277073
- [Derived] Makkar R, Butt J, Huang WY, McGlynn KA, Koshiol J, Pawlita M, Waterboer T, Freedman ND, Murphy G. Seropositivity for Helicobacter pylori and hepatobiliary cancers in the PLCO study. Br J Cancer. 2020 Sep;123(6):909-911. doi: 10.1038/s41416-020-0961-0. Epub 2020 Jun 29. PMID 32595210
- [Derived] Kunzmann AT, Coleman HG, Huang WY, Berndt SI. The association of lifetime alcohol use with mortality and cancer risk in older adults: A cohort study. PLoS Med. 2018 Jun 19;15(6):e1002585. doi: 10.1371/journal.pmed.1002585. eCollection 2018 Jun. PMID 29920516
- [Derived] Playdon MC, Ziegler RG, Sampson JN, Stolzenberg-Solomon R, Thompson HJ, Irwin ML, Mayne ST, Hoover RN, Moore SC. Nutritional metabolomics and breast cancer risk in a prospective study. Am J Clin Nutr. 2017 Aug;106(2):637-649. doi: 10.3945/ajcn.116.150912. Epub 2017 Jun 28. PMID 28659298
- [Derived] Piper MR, Freedman DM, Robien K, Kopp W, Rager H, Horst RL, Stolzenberg-Solomon RZ. Vitamin D-binding protein and pancreatic cancer: a nested case-control study. Am J Clin Nutr. 2015 Jun;101(6):1206-15. doi: 10.3945/ajcn.114.096016. Epub 2015 Apr 22. PMID 25904602